CLINICAL TRIAL: NCT04718155
Title: Could Early Atorvastatin Offer Anti Inflammatory Effects Upon Brain in Traumatic Head Injury? a Randomized Double-blind Clinical Trial
Brief Title: Could Early Atorvastatin Offer Anti Inflammatory Effects Upon Brain in Traumatic Head Injury?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB5566000
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; N-acetyl-aspartate
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- statin group (Active Comparator): will receive atorvastatin for 48 hours
  Interventions: Drug: Atorvastatin
- control (Placebo Comparator): will receive placebo tablets for 48 hours
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Atorvastatin — will receive 40 mg atrorvastatin 2 days
  Arms: statin group
Other: placebo — will receive 40 mg placebo 2 days
  Arms: control

SUMMARY:
3-Hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors, known as statins, are widely used to reduce levels of low-density lipoprotein-cholesterol. As lipid-lowering drugs, statins exert neuroprotective effects on ischemic stroke. this study will investigate whether the protective effect of statins is mediated by their ability to impact inflammation and oxygen free radical levels in cerebral ischemia/reperfusion injury.

Could Statins affect the neuroinflamation which occurs after traumatic brain injury?

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is one of the most common and financially devastating health problems in our society. Once the acute care period has ended, many TBI patients are left with motor, cognitive, or emotional dysfunction as a result of their injury. The treatment of TBI remains largely supportive, directed toward management of cerebral edema and intracranial hypertension via temporizing measures, such as administration of osmotic agents, hyperventilation, and ventricular drainage. None of these interventions have been definitively demonstrated to improve long-term functional outcome. The failure of preclinical therapies to translate into clinical benefit may derive from the heterogeneity of TBI pathology, which includes diffuse axonal injury, cerebral contusion, intracerebral hemorrhage (ICH), subarachnoid hemorrhage (SAH), and extra parenchymal hemorrhage. These primary insults are exacerbated by a secondary neuroinflammatory cascade of cerebral hypoperfusion and ischemia, oxidative stress, cerebral edema, and intracranial hypertension. There are a series of reactions following cerebral ischemia/reperfusion, such as inflammation and an increase in free radicals, which may trigger secondary injury in ischemic tissue. Indeed, the inhibition of inflammation reduces tissue damage in ischemia. Thus, understanding the roles of inflammation and free radicals in ischemia/reperfusion injury is therefore of great importance.

3-Hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors, known as statins, are widely used to reduce levels of low-density lipoprotein-cholesterol. As lipid-lowering drugs, statins exert neuroprotective effects on ischemic stroke. In this study, teh study will investigate whether the protective effect of statins is mediated by their ability to impact inflammation and oxygen free radical levels in cerebral ischemia/reperfusion injury. Statins have been shown to reduce morbidity in patients who did not have high serum cholesterol or cardiovascular disease but did have evidence of systemic inflammation. Statins have strong efficacy on modulation of inflammatory responses. conditions where statins have been found to have a positive effect on disease progression or mortality are primarily dependent on leucocyte accumulation. Statins may thus promote the timely resolution of the inflammatory response, preventing persistence of inflammation and resultant pathology.

Magnetic resonance spectroscopy (MRS) allows for measurement of metabolites that are undetectable by conventional neuroimaging thereby holding potential to identify traumatic brain injury patients that could benefit from specific neuropsychiatric and cognitive rehabilitation . Brain energy metabolism is altered after TBI due to posttraumatic inflammation and ischemia with mitochondrial dysfunction and loss of neuronal integrity with increased cell membrane turnover. MRS is an MRI technique that can detect nuclei with spins such as 1H, an abundant by-product of cellular respiration and brain tissue metabolites. As a noninvasive and safe technique, MRS is available on clinical MR scanners (1.5 and 3.0 T) without ionizing radiation [15]. This method holds the potential to identify compromised brain metabolism, but evidence after traumatic brain injury is rare .

ELIGIBILITY:
Inclusion Criteria:

- adult

* traumatic brain injury mild to moderate

Exclusion Criteria:

* immunotherapey
* diabetic
* previous CNs dysfunction

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
brain magnetic resonance spectroscopy | first 48 hours
  presence or absence of abnormal metabolites seen by magnetic resonance spectroscopy

SECONDARY OUTCOMES:
ICU stay | first 30 days
  days of ICU stay

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt